CLINICAL TRIAL: NCT06432075
Title: Single Arm Clinical Prospective Study of Neoantigen Reactive T Cells (NRTs) in the Treatment of Chinese Patients With Advanced Gastric Cancer
Brief Title: Neoantigen Reactive T Cells c for Chinese Patients With Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Shen Xian, Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neoantigen T Cells
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Advanced Gastric Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen Reactive T Cells (Experimental): Peripheral blood lymphocytes will be collected and neoantigen reactive T cells(NRTs) will be generated in the laboratory;nab-paclitaxel 100-200mg/m2/D will be i.v. for 7 days before cell infusion; Cyclophosphamide 300mg/m2/D will be i.v. for 2 and 3 days before cell infusion; NRTs 0.5~1 x 10^10, will be i.v.Q3 weeks for total 4 doses;Interleukin-2 (IL-2) will be continuous intravenous infused since the first day of the cell infusion for 5 consecutive days, 1000,000 international unit per day.All Patients will receive a total of 4 cycles of treatment.
  Interventions: Biological: Neoantigen Reactive T Cells(NRTs)

INTERVENTIONS:
Biological: Neoantigen Reactive T Cells(NRTs) — Neoantigen Reactive T Cells in an expected volume of 100 milliliter（mL） will be given by intravenous injection over 2-10 minutes through either a peripheral or a central line.

SUMMARY:
The purpose of this study is to see the safety and efficient of neoantigen reactive T cells (NRTs) in the treatment of Chinese patients with advanced gastric cancer.

DETAILED DESCRIPTION:
The tumor-specific "none-self" immunogenic neoantigens encoded by either viral genes or somatic mutation genes, possess the potential to induce specific anti-cancer immunity, including cellular and humoral immune responses. Today, numerous clinical trials demonstrate that although these "none-self" antigens initiate the antigen-specific immunoglobulin G antibodies and cluster of differentiation 4（CD4）+/cluster of differentiation 8（CD8）+T-cells response, not all of them show a clinical benefit in the response rate, progression-free survival or overall survival.Personalized cell therapy maybe own a breakthrough in the treatment of those gastric cancer patients without standard options.The investigators' center has successfully established a new method for preparing personalized neoantigen reactive T cells(NRTS) for adoptive cell therapy(ACT). Today, the investigators will carry out a single arm clinical prospective study of NRTs for the treatment of Chinese patients with advanced gastric cancer. Participants are assigned to receive 4 circles of cell therapy, and IL-2 continuous intravenous infusion（CIV） will also be given for 5 consecutive days after each time's cell infusion. The safety and clinical response rate（RR） are evaluated. Biomarkers and immunological markers are also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join the study and sign the informed consent;
2. Age: 18-75 years old, male or female;
3. Subjects with advanced gastric cancer who had received systematic standard treatment before enrollment and had no effective treatment at present. (Note: The effective treatment means refer to the latest version of the "Gastric Cancer Diagnosis and Treatment Guide" issued by China's "Chinese Clinical Oncology Society".) ;
4. Have at least one measurable lesion according to imRECIST evaluation criteria;
5. Expected survival ≥5 months (starting from the collection of tissue samples for sequencing);
6. The Eastern Cancer Consortium (ECOG) score was 0 or 1 or 2;
7. The following hematological indicators should be met: neutrophil count ≥ 1.5×109/L; Hemoglobin ≥ 10.0 g/dL; Platelet count ≥ 50×109/L;
8. The following biochemical indicators should be met: total bilirubin ≤2.0× upper limit of normal value (ULN); AST and ALT ≤2.0×ULN; Serum creatinine ≤1.5×ULN.
9. Before lymphocyte clearance preadministration: 1) any chemotherapy, small molecule targeted drugs and other antitumor therapy received have passed the 3-week washout period, and the toxic side effects have returned to grade 1 or lower (excluding hair loss, vitiligo and other events as determined by the investigator to be tolerated); 2) If surgical treatment is performed within 3 weeks, toxicity has returned to grade 1 or lower; 3) The immunotoxicity of major organs has returned to grade 1 or lower after receiving any antibody drug treatment, and the washout period of PD-1 antibodies has reached 6 weeks, and CTLA-4 antibodies and other antibodies have passed the washout period of 4 weeks.

Exclusion Criteria:

1. Subjects infected with HBV, HCV, HIV, syphilis and tuberculosis;
2. Uncontrolled coronary artery disease or asthma, uncontrolled cerebrovascular disease or what the investigator considers Other diseases not included in the group;
3. Patients with a history of bone marrow or organ transplantation; Patients with coagulation dysfunction;
4. Patients with immune deficiency diseases or autoimmune diseases who are treated with immunosuppressive drugs;
5. Central nervous system (CNS) metastatic and/or cancerous meningitis;
6. People who may be allergic to immunotherapy;
7. Drug abuse, clinical or psychological or social factors that affect informed consent or the conduct of the study;
8. Pregnant and lactating women;
9. Participating in other clinical trials;
10. An uncertainty that the investigator believes has an impact on the subject's safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | up to 6 months
  using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients

SECONDARY OUTCOMES:
Response Rate | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  Response Rate（RR）will be evaluated according Response Evaluation Criteria in Solid Tumors
Progression free survival (PFS) | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  the duration of progression free survival is measured from the time of treatment to the first date that recurrent or progressive disease or for any reason of death is objectively documented.

OTHER OUTCOMES:
Overall Survival (OS) | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  the duration is measured from the time of treatment to the time of death
Interferon-gama change of PBMC cells in the peripheral blood stimulated by tumor antigens | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  T cells in the peripheral blood stimulated by tumor antigens for 24 hr，and then Interferon-gama secretion is measured

IPD SHARING:
Plan to Share IPD: No
Publications